CLINICAL TRIAL: NCT05896436
Title: Emotion Focused Therapy for Depression and Anxiety Among Competitive Athletes - A Feasibility Study
Brief Title: Emotion Focused Therapy for Competitive Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Katherine Tamminen, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00044207; 430-2022-00033 (Other Grant/Funding Number: Social Sciences and Humanities Research Council of Canada)
Record Dates: First submitted 2023-04-06; First posted 2023-06-09 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Emotion-Focused Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Focused Therapy (Experimental): Participants will receive 12 weekly 1-hour sessions of Emotion Focused Therapy with a trained student therapist.
  Interventions: Behavioral: Emotion Focused Therapy
- Wait list control (No Intervention): No intervention; waitlist control group will receive intervention once the data collection during the intervention period has concluded.

INTERVENTIONS:
Behavioral: Emotion Focused Therapy — 12 sessions of Emotion Focused Therapy (EFT). The focus in EFT is to promote the individual's experiencing and facilitate participants' self-disclosure and openness to their own experience, rather than the therapist's agenda or techniques. Key processes within EFT include helping people overcome their avoidance of emotion, maintaining a collaborative focus on emotions, and exploring emotions in therapy.
  Arms: Emotion Focused Therapy

SUMMARY:
This project will be a pilot study to test the feasibility of using Emotion Focused Therapy (EFT) among competitive athletes experiencing mild-to-moderate depression or anxiety. To test whether the intervention works, the researchers will assess athletes' emotion dysregulation, symptoms of mood disorders (anxiety and depression), sport-related distress, subjective performance satisfaction, and well-being. In addition to assessing athlete outcomes, key aspects to be examined in the pilot study include the recruitment and randomization procedures, informed consent procedures, data collection tools, implementation of the intervention, and retention of participants. Feasibility will be assessed by recruitment (willingness to be randomized, number of eligible participants in the recruitment process). Retention will be assessed by the number of athletes who continue or discontinue attendance. Participants' experiences in the intervention will be assessed via qualitative interviews to gain in-depth information about their perceptions of the intervention.

DETAILED DESCRIPTION:
This project will be a pilot study to test the feasibility of using Emotion Focused Therapy (EFT) among 24 competitive athletes over the age of 18 in Ontario. Athletes will be screened and allocated to receive 12 weekly one-hour sessions of Emotion Focused Therapy, or they will be allocated to a wait-list control group.

Screening: Participants interested in the study can contact the study coordinator, who will provide them with information about the study and conduct an initial screening process to ask them their age, competitive level, and province of residence. Athletes who are under the age of 18, not participating in competitive sport, or not living in Ontario will not be eligible to participate in the study; these athletes will be provided with community mental health support information if they would like to seek other options for mental health support. Athletes who are over the age of 18, participating in competitive sport, and living in Ontario will be provided with information about the study and the study coordinator will review the information letter verbally with them and answer any questions they have about the study. If they are interested in participating, they will be sent the baseline survey measures (to be completed online) and responses will be screened to determine whether the intervention will be appropriate for them.

Measures: The measures include a demographics form and the primary and secondary outcome measures. After completing these measures online, the study coordinator will score and screen the measures to determine the participant's eligibility to be allocated to the study. Athletes whose scores indicate severe levels of anxiety or depression, or who indicate a high likelihood of an eating disorder, will be referred for immediate treatment and will be not be eligible for the study from the study. Athletes who indicate low levels of depression or anxiety will not be eligible for the study and provided with information about mental health support services. Participants will be randomly allocated to the intervention condition or a wait-list control group; once assigned to the intervention group, participants will also be assigned on a rotating basis to the three student therapists delivering the intervention. The study coordinator will electronically randomize participants to the intervention or wait-list control group. Participants will not be blinded to their group allocation.

Intervention: The Emotion Focused Therapy (EFT) intervention is a process-experiential approach to psychotherapy that is grounded in humanistic approaches to therapy. EFT focuses on promoting client experiencing and being nondirective; that is, the therapist emphasizes facilitating clients' self-disclosure and openness to their own experience, rather than the therapist's agenda or techniques. Key processes within EFT include helping people overcome their avoidance of emotion, maintaining a collaborative focus on emotions, and exploring emotions in therapy. The role of the therapist in EFT is considered as an 'emotion coach' and guides the processing of emotions. While there is no set schedule for the sessions, common tasks that may arise in the course of therapy include developing a therapeutic alliance with the athlete; increasing awareness and attention to emotions; increasing capacity tolerance of emotional arousal; validation of emotional experience; evocation and exploration of emotions; and transformation of emotions (helping athlete develop new emotional responses and making sense of experiences, validating new feelings and an emerging sense of self).

Survey Timing: Athletes will complete baseline questionnaires before randomization, at postintervention, and at follow-up one month later.

Post-Intervention Interview: Participants will be invited to take part in an online interview following the completion of the intervention and after completing the final survey in the study. Participants will be asked about their experiences during the intervention and their experiences of receiving Emotion Focused Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 and capable of consenting to participate in the study
* Participating in competitive sport (highly trained/national level or above); athletes may be participating in any able-bodied or para-sport.
* Speak and comprehend English
* Meet criteria for mild-to-moderate depression or anxiety
* Reside in Ontario
* Not currently receiving psychotherapy

Exclusion Criteria:

* Athletes under the age of 18 who are not able to provide informed consent to participate in the study
* Athletes participating in recreational sport
* Athletes who meet criteria for high risk of eating disorder
* Athletes who meet criteria for severe depression or anxiety
* Athletes who do not live in Ontario
* Athletes indicating low levels of depression or anxiety
* Athletes who are currently receiving psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline score in depressive symptoms | At 12 weeks or immediately after termination of intervention, if terminated earlier than 12 sessions.
  Depression will be assessed using the Patient Health Questionnaire (PHQ-9), which is a 9-item, self-report questionnaire designed to assess the participant's depression levels during the past 2 weeks. The PHQ-9 utilizes a 4-point scale (0= not at all, 3= nearly every day). Scores are totaled and presented from 0 to 27. Scores of 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe, and severe depression, respectively.
Change from baseline score in anxiety symptoms | At 12 weeks or immediately after termination of intervention, if terminated earlier than 12 sessions.
  Anxiety will be assessed with the Generalized Anxiety Disorder Scale (GAD-7), which is a 7-item, self-report anxiety questionnaire designed to assess the participant's anxiety levels during the past 2 weeks. The GAD-7 utilizes a 4-point scale (0= not at all, 3= nearly every day). Scores are totaled and presented from 0 to 21. Scores of 5, 10, and 15 represent cut-off points for mild, moderate, and severe anxiety, respectively.

SECONDARY OUTCOMES:
Change from baseline score in Emotion Dysregulation | At 12 weeks or immediately after termination of intervention, if terminated earlier than 12 sessions.
  Emotion Dysregulation measured using the Difficulties in Emotion Regulation Scale. Items are rated on a scale of 1 (almost never [0-10%]) to 5 (almost always [91-100%]). Scores are summed (scores ranging from 36-180) with higher scores indicate more difficulty in emotion regulation.
Change from baseline score in alexithymia | At 12 weeks or immediately after termination of intervention, if terminated earlier than 12 sessions.
  Alexithymia measured using the Toronto Alexithymia Scale-20. Items are rated on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). The total score can be used from the three subscales, or the sum of each subscale score can be used; for the present study only the subscales related to difficulty in identifying feelings and difficulty in describing feelings will be used; higher scores indicate greater degree of difficulty in identifying feelings and describing feelings.
Change in baseline score for Sport Related Distress - Athlete Psychological Strain | At 12 weeks or immediately after termination of intervention, if terminated earlier than 12 sessions.
  Sport-Related Distress will be measured using the Athlete Psychological Strain Questionnaire (APSQ). The APSQ utilizes a 5-point scale (1 = "None of the time"; 5 = "All of the time"). Scores are totaled and presented from 10 to 50 with a higher score indicating more psychological strain.
Changes in baseline score for Sport Related Distress - Sport Psychology Outcomes | At 12 weeks or immediately after termination of intervention, if terminated earlier than 12 sessions.
  Sport-Related Distress will be measured using the Sport Psychology Outcomes and Research Tool (SPORT). The SPORT utilizes a 5-point scale (1= Strongly Agree, 5= Strongly Disagree) where statements 16 and 17 are reverse coded, and lower scores reflect better functioning.

OTHER OUTCOMES:
Client-Therapist Working Alliance | Working alliance will be assessed at 4 weeks, 8 weeks, and 12 weeks during the intervention.
  Therapist Working Alliance will be measured using The Working Alliance Inventory-Short Revised, which is a 12-item measure of three factors reflecting agreement on goals of the therapy (Goal Scale: 4 items), agreement that the tasks of the therapy will address the problems the athlete is experiencing (Task Scale: 4 items), and the quality of the interpersonal bond between the athlete and the therapist (Bond Scale: 4 items). Items at rated on a 5-point scale from 1 (never) to 5 (always) and higher scores reflect a better working alliance.
Athletes' experiences of participating in psychotherapy | After conclusion of intervention (one-month follow up).
  Perceptions about experiences with the intervention will be explored using qualitative interviews with athletes at post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tamminen, PhD, Principal Investigator — University of Toronto
Locations (1):
- Faculty of Kinesiology and Physical Education, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study will be stored in a non-publicly available repository (Dataverse: https://borealisdata.ca/dataverse/toronto). De-identified survey data and interview transcripts will be stored indefinitely in an online repository (Dataverse). Researchers wishing to access the data for research purposes/secondary analyses will require ethical approval from a recognized research ethics board and submit a request for access to the data from the lead investigator. No personally-identifying data will be stored, only variable data and results. Participants will be asked to provide consent to store their data for future research purposes.
Supporting Information: Study Protocol, ICF
Time Frame: Intention to publish date: 30/06/2025
Access Criteria: Researchers wishing to access the data for research purposes/secondary analyses will require ethical approval from a recognized research ethics board and submit a request for access to the data from the lead investigator.

DOCUMENTS (1):
  • Informed Consent Form (2023-03-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT05896436/ICF_000.pdf